CLINICAL TRIAL: NCT01132469
Title: Long-term Follow-up After Endoscopic Submucosal Dissection for Early Gastric Cancer
Brief Title: Efficacy and Safety Study of Endoscopic Submucosal Dissection for Early Gastric Cancer
Acronym: ESD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Eunhee Shin/General Manager of Pragmatic Clinical Trials Team, National Evidence-based Healthcare Collaborating Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA09-003
Record Dates: First submitted 2010-05-24; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Endoscopic Submucosal Dissection; Early Gastric Cancer; Multi-center, Single-arm Clinical Trial; Historical Control Group; Quality of Life and Cost Analysis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopic Submucosal Dissection (Experimental): Single-arm for ESD procedure and retrospective surgical procedure(Laparoscopy, Open surgery)data collection
  Interventions: Procedure: Endoscopic Submucosal Dissection

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — 5-years follow-up after Endoscopic Submucosal Dissection

SUMMARY:
The purpose of this study is to evaluate the safety and clinical effectiveness of ESD(Endoscopic Submucosal Dissection) for early gastric cancer analyzing short-term and long-term results of endoscopic treatment.

DETAILED DESCRIPTION:
Traditionally open-gastrectomy is the standard treatment for gastric cancer without distant metastasis, but high mortality and morbidity, the intense weight loss, food intake difficulties after surgery are fraught, including problems with the drawback of significantly degrading the quality of life. Therefore, a lot of effort to seek the more simple treatment than open gastrectomy has been made, recently the endoscopic treatment for early gastric cancer is the most widely used treatment.

This single-arm, multi-center study enroll early gastric cancer patients after ESD compared with the retrospective control(surgical treatment) group considering the unreality of the randomized clinical trials. In addition, the quality of life assessment by the EORTC C30/STO22 tools before and after ESD procedure in enrolled patients will be performed and the direct cost analysis also will be conducted.

ELIGIBILITY:
1. ESD GROUP

   Inclusion Criteria:
   * Korean people aged >=20 years
   * Endoscopic Grossly the lesion diameter ≤ 3cm
   * Endoscopic biopsy results: Well-differentiated and moderately differentiated adenocarcinoma
   * No ulcers in lesions
   * Endoscopic biopsy results: In case of gastric cancer, no metastasis in CT test performed before ESD procedure

   Exclusion Criteria:
   * Subject with history of malignant disease in other organs
   * Subject with history of stomach surgery due to peptic ulceration etc.
   * As the cases of an absolute contraindication of general anesthesia; Subject with chronic liver disease over Child score B, Subject with chronic Renal Disease requiring hemodialysis or peritoneal dialysis, Subject with heart failure more than Ⅲ score according to New York Heart Association Classification, Subject with severe systemic diseases such as respiratory disease
   * Subject with Bleeding tendency
   * Pregnant woman or woman with possibility of pregnancy
   * Subject who cann't be obtained informed consent
   * Subject who is unable to follow up for any other reason
2. Surgery Group(Retrospective data collection)

Inclusion Criteria:

* Subject with gastric laparoscopy or open-surgery for treatment early gastric cancer during 2002.1.1 ~2004. 12. 31
* Korean people aged >=20 years
* Early gastric cancer confirmed by pathology during gastric surgery; Gastric cancer confirmed to the mucosal or submucosal regardless of lymph node metastasis
* No history of malignant disease in other organs
* No history of stomach surgery due to peptic ulceration etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1158 (Estimated)
Dates: Start 2010-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
5-year disease(gastric cancer)-free survival rate after ESD procedure | 5 years after ESD

SECONDARY OUTCOMES:
Short-term result(Histological complete resection,complication) | within the first 7 days after ESD
The incidence of reoccurrence and Ectopic foci | within the first 7 days and 3months, 6months, 1year, 2years, 3years, 4years and 5years after ESD
The quality of life after ESD | before and 7 days, 3months, 6months after ESD
The costs of ESD | From the admission to discharge
The safety of ESD procedure | within the 7 days, 3months, 6months, 1year, 2years, 3years, 4years and 5years after ESD

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Yong Seol, M.D., Principal Investigator — Inje University College of Medicine
Locations (1):
- Inje University Busan Baik Hospital and 10 other institutes, Busan, South Korea